CLINICAL TRIAL: NCT04698434
Title: The Best Dose of Esketamine for Day Surgery of Pediatric Circumcision
Brief Title: The Best Dose of Esketamine for Day Surgery of Pediatric Circumcision Pediatric Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Ma Hong, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y015
Record Dates: First submitted 2020-07-31; First posted 2021-01-06 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Phimosis
Keywords: Esketamine; Sevoflurane; Children; circumcise
MeSH Terms: conditions — Phimosis | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: children who underwent day surgery of pediatric circumcision were randomly divided into 3 groups according to the random number table method:0.5mg/kg esketamine group (Group A), 0.75mg/kg esketamine group (Group B) and 1.0mg/kg of esketamine group (Group C), with 30 people in each group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.5mg/kg esketamine group (Active Comparator): 0.5mg/kg esketamine group will be given a single intravenous 0.5mg/kg esketamine
  Interventions: Drug: Esketamine
- .75mg/kg esketamine group (Active Comparator): 0.75mg/kg esketamine groupwill be given a single intravenous 0.75mg/kg esketamine
  Interventions: Drug: Esketamine
- 1.0mg/kg esketamine group (Active Comparator): 1.0mg/kg esketamine group will be given a single intravenous 1.5mg/kg esketamine
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — each group was given a single intravenous dose of the corresponding esketamine.

SUMMARY:
In recent years, daytime operation has been developed gradually in China. Circumcision in children is a common type of daytime operation. The nature of the operation and the object of the operation determine that the anesthetic drugs used should induce fast, wake up quickly and recover in a high quality.

Esketamine is an S-enantiomer of ketamine, which is newly marketed in China. Compared with ketamine, it has stronger effect on NMDA receptor, and its sedative effect is about twice as high. The occurrence frequency of respiratory depression and hypotension is lower than that of other anesthetics and analgesics, which can provide good analgesic and sedative effect for surgical anesthesia.

In clinical practice, ketamine combined with sevoflurane has been widely used in children's microsurgery, but there has been no report on Esketamine combined with sevoflurane anesthesia.

In order to find out the best combined dose, this paper compares the single administration of three different doses of esketamine combined with sevoflurane anesthesia in the circumcision of children.

DETAILED DESCRIPTION:
To investigate the optimal dose of esketamine combined with sevoflurane for pediatric circumcision. Methods children who underwent day surgery of pediatric circumcision were randomly divided into 3 groups according to the random number table method:0.5mg/kg esketamine group (Group A), 0.75mg/kg esketamine group (Group B) and 1.0mg/kg of esketamine group (Group C), with 30 people in each group. mask inhalation of sevoflurane anesthesia, each group was given a single intravenous dose of the corresponding esketamine. Heart rate (HR), mean arterial pressure (MAP), pulse oxygen saturation (SpO2) and respiratory rate (RR) were recorded at room entry (T0), intravenous ketamine administration (T1), operation initiation (T2), intraoperative central ligation (T3) and operation completion (T4).The number and total amount of ketamine added intraoperatively were recorded. Duration of operation, time to open eyes and time to answer were recorded. The Eastern Ontario Children's Hospital pain Score (CHEOPS score) and the modified Bieri pain score were recorded when awake, 2 hours and 6 hours postoperatie. MOAA/S score was recorded at 15, 30 and 60min after surgery. Intraoperative and post-operative adverse reactions were recorded, including hypersensitivity, agitation, nausea and vomiting, dizziness, diplopia, etc.

ELIGIBILITY:
Inclusion Criteria:

* phimosis

Exclusion Criteria:

* cardiopathy
* asthma
* dysgnosia
* surdimutism
* hepatopathy or nephropathy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
recovery time | up to 2 hour
  the time from stopping sevoflurane to resuscitation

SECONDARY OUTCOMES:
CHEOPS score | up to 6 hours
  The Eastern Ontario Children's Hospital Pain Score (CHEOPS score) at the time of 2h and 6h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sun Ji Hong, bachelor, Study Chair — Yangzhou University
Locations (1):
- Affiliated hospital of yangzhou university, Yangzhou, Jiangsu, China